CLINICAL TRIAL: NCT05168046
Title: Pilot Study of the Ambulatory Monitoring Evaluation of a Mindfulness Meditation Programme in Parkinsonian Tremor
Brief Title: Mindfulness-based Intervention for People With Parkinsonian Tremor
Acronym: MEDITAPARK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Institut National de Recherche en Informatique et en Automatique (Other); Université Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RECHMPL20_0321
Record Dates: First submitted 2021-10-29; First posted 2021-12-23 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Parkinson Disease; Rest Tremor
Keywords: parkinson disease; rest tremor; mindfulness based intervention; sensors; embrassment
MeSH Terms: conditions — Parkinson Disease; Tremor | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Parkinson Mindfullness Based Stress Reduction (Experimental): Patients who have an assessment before and after a mindfulness based stress reduction intervention for 6 months
  Interventions: Behavioral: Mindfulness based stress reduction
- Parkinson controls (No Intervention): Patients who have an assessment before and after 6 monthswithout intervention

INTERVENTIONS:
Behavioral: Mindfulness based stress reduction — program of weekly mindfulness based stress reduction intervention during 2 months and practice during 3 months
  Arms: Parkinson Mindfullness Based Stress Reduction

SUMMARY:
Mindfulness meditation is an approach that has shown interest in treatment of anxiety in Parkinson's disease. This pilot study aims to assess a more specific effect on tremor using Essential Tremor Embarrassment Assessment and inertial sensors allowing monitoring during sessions and in daily life. This study will focus on 20 patients (10 with and without Mindfulness based intervention and will aim to develop the interface and demonstrate proof of concept before setting up a controlled study

DETAILED DESCRIPTION:
Methodology: Randomized, pilot study comparing 2 parallel arms (Mindfullness group versus group with routine care).

Number of patients:20

Patient selection: patients with severe rest tremor

Duration of project: 12 months

Schedule visit: 4 visits in 6 months

ELIGIBILITY:
Inclusion Criteria:

* Parkinson disease
* Hoehn st and yahr stage <or = 3
* Age between 35 and 85 years old
* Treatment stabilized for at least 3 months
* Disturbing parkinsonian tremor of the upper limb (item MDS -UPDRS 2.10> 1) and lasting 2 to 6 hours per day
* patients with internet access

Exclusion Criteria:

* Presence of disturbing dyskinetic movements (Item MDS-UPDRS4.2> 1)
* Patient who has already practiced meditation in the last 5 years
* Untreated major depressive episode
* Hallucinations (Item MDS-UPDRS1.2> 1))
* Psychotic disorders - Confusional syndrome
* presence of signs in favor of an atypical parkinsonian syndrome (oculomotor impairment, early falls, hallucinations, MoCA <20, early dysautonomia)
* adult protected by law (guardianship, curatorship or under legal protection)

  * deprivation of liberty by judicial or administrative decision
  * high probability of non-compliance with the protocol or abandonment during the study
* refusal to sign informed consent
* Pregnant or breastfeeding woman
* Lack of social coverage.

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2024-10-20 (Actual); Study Completion 2024-10-20 (Actual)

PRIMARY OUTCOMES:
Essential Tremor Embarrassment Assessment score | Month 6 (M6)
  Essential Tremor Embarassment Assessment scale, ETEA : this scale is a self questionnaire made up of 14 items (0 to 5, 5 = worst embarrassment)

SECONDARY OUTCOMES:
duration of tremor assessed by agenda | Day 0 (inclusion), Month 3 (M3)
  Weekly cumulative time differences of tremor periods on Hauser's modified auto-diary (2000)
duration of tremor assessed by sensors monitoring | Day 0 (inclusion), Month 3 (M3)
  Weekly cumulative time differences of tremor periods recorded with the connected watch
feasability of the study : number of patients enrolled | Month 6 (M6)
  - Proportion of patients included among screened patients
feasability of the study : number of patients ended the study | Month 6 (M6)
  - Proportion of patients who completed the meditation program
feasability of the study : hours of recording of the tremor | Month 6 (M6)
  - Proportion of hours of recording of the tremor compared to the planned duration
feasability of the study : tolerance | Month 6 (M6)
  Tolerance to the meditation program assessed with a 10-point Likert scale
feasability of the study : COREQ 1 | Month 6 (M6)
  - Focus Groups Consolidated Criteria for Reporting on Qualitative Studies (COREQ) 1
Severity tremor index assessed by sensors monitoring | Month 3 (M3)
  Differences in the Severity tremor index (mean amplitude of the tremor measured by the smartwatch)
Quality of life : Parkinson Disease Questionnaire 39 (PDQ39) scale | Month 6 (M6)
  The PDQ39 scale is a self questionnaire made up of 39 items exploring 8 dimensions (mobility, daily activities, emotionnal well-being, psychological incomfort, social support, cogntive disorders, communication, physical incomfort).
  Description: Parkinson Disease Questionnaire 39 Quality of Life Score (PDQ39) (Auquier et al., 2002) - The PDQ-39 is a self-administered health-related Quality of Life (QOLL) instrument made up of 39 items exploring 8 dimensions (mobility , activity of daily living, emotional well-being, psychological discomfort, social support, cognitive disorders, communication, physical discomfort)
Quality of life : Hamilton anxiety and depression scale (HADS) | Month 6 (M6)
  Depression score: Hamilton Anxiety and Depression Scale (Leentjeens, 2011) - This questionnaire assesses the presence and severity of anxiety and depressive symptoms.
  14 questions, answers between 0 and 3, total score between 0 and 42, 42 is the worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Montpellier University Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: No